CLINICAL TRIAL: NCT07327307
Title: A Real-World Registry Study to Evaluate Clinical Protection Outcomes Following Post-Exposure Prophylaxis With Zamerovimab and Mazorelvimab Injection in Combination With Rabies Vaccine in Pediatric With Category III Rabies Exposure
Brief Title: Real World Evidence Study of SYN023 in Children Exposed to Rabies
Status: Recruiting | Type: Observational
Sponsor: Synermore Biologics (Suzhou) Co., Ltd. (Industry)
Collaborators: Peking University First Hospital (Other); Shenzhen Second People's Hospital (Other); Hunan Provincial People's Hospital (Other); The University of Hong Kong-Shenzhen Hospital (Other); University of South China Affiliated Nanhua Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: SYN023-008
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Rabies Post-exposure Prophylaxis
Keywords: rabies; SYN023; pediatric
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SYN023 combined with rabies vaccine
- Other rabies passive immunization products combined with rabies vaccine

SUMMARY:
This observational study is an open-label, prospective, multi-center design. The goal is to evaluate the long-term clinical survival outcomes at 3 months and 1 year in individuals under 18 years of age with WHO Category III rabies exposure who have received real-world Post-Exposure Prophylaxis (PEP) with Zamerovimab and Mazorelvimab Injection / other passive immunization products combined with the rabies vaccine.

Participants will: (1) Have their clinical protection outcomes (rabies-free survival status) registered and evaluated on Day 90 and Day 365. (2) Have the option to provide a blood sample on Day 7 for Rabies Virus Neutralizing Antibody (RVNA) testing. (3) Have all adverse events (within 42 days) and all serious adverse events (within 126 days) after PEP administration collected and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age under 18 years on the day of enrollment, regardless of gender, and able to provide legal proof of identity;
2. Individuals with WHO Category III rabies exposure, and the time from exposure to the initiation of Post-Exposure Prophylaxis (PEP) is <7 days;
3. Have completed standardized wound management, injection of Zamerovimab and Mazorelvimab Injection /other passive immunization products, and the first dose of rabies vaccination within 24 hours prior to screening;
4. The volunteer's guardian voluntarily agrees to their participation in the study and signs the informed consent form. Specifically: for volunteers under 8 years old, the guardian signs the informed consent form with the child's assent fully respected; for volunteers aged 8-17, the guardian signs the informed consent form, and the minor volunteer signs the minor assent form;
5. Willing and able to comply with all study procedures, and is expected to be able to complete the full course of rabies vaccination and the 1-year follow-up as required (with no plans for long-term absence or relocation from the study area).

Exclusion Criteria:

1. Based on inquiry, besides the current Category III rabies exposure, there is a history of bites by dogs, cats, mongooses, foxes, ferrets, skunks, bats, or raccoons within the past year;
2. Other conditions considered by the investigator as unsuitable for participation in this study.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Individuals under 18 years of age with category III rabies exposure who have received post-exposure prophylaxis (PEP) with Zamerovimab and Mazorelvimab Injection /other passive immunization products combined rabies vaccine in the real world
Sampling Method: Non-Probability Sample
Enrollment: 232 (Estimated)
Dates: Start 2025-08-02 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rabies-free survival rate | 3 months and 1 year
  WHO's Classification of Rabies Cases:
  Suspected case: refers to a case that satisfies the definition of clinical case; Probable case: refers to a suspected case with a reliable medical history of contact with any suspected animal infected with the rabies virus; Confirmed case: refers to a suspected or probable case that is proved to be infected based on the lab test result.

SECONDARY OUTCOMES:
Incidence of adverse reactions and adverse events | 42 days
Incidence of serious adverse reactions and serious adverse events | 126 days
Rabies Virus Neutralizing Activity (RVNA) of Geometric Mean Concentration (GMC) | Day 7
Percentage of Participants With Rabies Virus Neutralizing Activity (RVNA) ≥0.5 IU/mL | Day 7

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Shenzhen second people's hospital, Shenzhen, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Affiliated Nanhua Hospital, University of South China, Hengyang, Hunan
  - Jiangxi Provincial Chest Hospital, Nanchang, Jiangxi